CLINICAL TRIAL: NCT00498173
Title: Targeted Pharmacologic Interventions for Autism: A Double-Blind, Placebo-Controlled Trial of Atomoxetine in Children and Adolescents With Autism
Brief Title: Effectiveness of Atomoxetine in Treating ADHD Symptoms in Children and Adolescents With Autism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christopher John McDougle, M.D., Director, Lurie Center for Autism, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH077600 (NIH); R01MH077600 (NIH); DDTR B2-NDA (Other)
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Autism
Keywords: Autistic Disorder; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: At the end of the 8-week double-blind, placebo-controlled study, participants randomized to placebo who are not responders at the end of 8 weeks will be treated with atomoxetine for 8 weeks during an open-label trial. All participants who are rated "much improved" or "very much improved" on the CGI-I following treatment with atomoxetine (i.e., atomoxetine responders) during either the 8-week placebo-controlled trial or the 8-week open-label phase for placebo nonresponders will be eligible to enter the 10-month open-label extension phase of the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomoxetine (Experimental): Participants will receive flexibly dosed atomoxetine for 8 weeks. Dosage can be increased over the first 4 weeks of study participation and will then be held constant for the remainder of the 8-week trial.
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Participants will receive blinded, matched placebo for 8 weeks. Dosage can be increased over the first 4 weeks of study participation and will then be held constant for the remainder of the 8-week trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Available tablet strengths of atomoxetine: 5 mg, 10 mg, 25 mg, 40 mg. Week 1 participant takes 0.5 mg/kg/day, Week 2: 0.8 mg/kg/day, Week 3: 1.2 mg/kg/day. Potential exists for dose increase at Week 4 to 1.8 mg/kg/day based on clinical global impression-improvement rating at Week 4.
  Other Names: Strattera
  Arms: Atomoxetine
Drug: Placebo — Placebo tablets dosages: 5 mg, 10 mg, 25 mg, 40 mg.
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of atomoxetine in treating children with attention deficit hyperactivity disorder symptoms associated with autistic disorder, Asperger's syndrome, and pervasive developmental disorder, not otherwise specified.

DETAILED DESCRIPTION:
Autism is a developmental disorder that can cause severe and pervasive impairment in thinking, feeling, language, and the ability to relate to others. It is usually first diagnosed in early childhood. Children with autism demonstrate repetitive behaviors or interests and deficits in social interaction, verbal communication, and nonverbal communication. In addition, they often have unusual responses to sensory experiences, such as certain sounds or the way objects look. Some symptoms of attention deficit hyperactivity disorder (ADHD), such as inattention, hyperactivity, and impulsivity, are also associated with autism. Atomoxetine is a selective norepinephrine reuptake inhibitor that is used to treat ADHD. It works differently, however, than stimulant drugs and may help to reduce ADHD symptoms in children with autism. This study will evaluate the effectiveness of atomoxetine in treating children with ADHD symptoms associated with autism.

Potential participants will first attend a screening visit, which will include a psychiatric diagnostic interview, a practice session for swallowing pill capsules, a physical exam, an electrocardiogram (ECG), a blood test, and an assessment of pubertal stage. Females of childbearing age will also undergo a urine pregnancy test. In an initial double-blind study phase, eligible participants will be randomly assigned to receive either atomoxetine or placebo for 8 weeks. A baseline visit will include several rating scales, observations, and an interview to assess adaptive functioning. These measures and procedures will be used to keep track of symptoms, side effects, and behavior that could change during the study. Children who are assigned to placebo and do not notice an improvement in their ADHD symptoms will be given the opportunity to receive atomoxetine at the end of 8 weeks. Study visits will occur once a week for 4 weeks, and then every other week for the remainder of the 8 weeks. During these visits, many of the baseline questionnaires and interviews will be repeated. At the Week 8 visit, the physical exam, ECG, blood tests, and some baseline questionnaires will also be repeated. All children who respond well to atomoxetine may continue taking the drug for an additional 10 months. During this time, participants will report to the clinic once a month for the first 4 months, then once at the end of 7 months, and finally once at the end of 10 months. The same measures and procedures that were done during the 8-week phase will be done during the 10-month phase of this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an autism spectrum disorder (autistic disorder, Asperger's syndrome, and pervasive developmental disorder, not otherwise specified).
* Significant hyperactivity, inattention, or impulsivity as determined by a score on an investigator-administered ADHD Rating Scale (ADHDRS)-Home Version that is at least 1.5 standard deviations above the mean for age and sex
* Parent/caregiver's primary complaint about the child is inattention, hyperactivity, and/or impulsivity ("ADHD" symptoms)
* Symptoms present for 6 months prior to study entry
* Psychotropic drug-free for at least 2 weeks prior to starting study medication. This drug-free period will be 5 weeks for fluoxetine (Prozac).

Exclusion Criteria:

* Weighs less than 15 kg (about 33 pounds)
* Any another psychiatric disorder that may require a different treatment, including psychotic disorders, major affective disorders, obsessive-compulsive disorder, panic disorder, or substance-related disorders
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of Rett's disorder or childhood disintegrative disorder
* Presence of extreme aggression or self-injury
* Currently taking an effective psychotropic drug
* Currently using other medications that may be unsafe to take with atomoxetine (e.g., potent CYP 2D6 inhibitors, intravenous albuterol, monoamine oxidase inhibitors[MAO])
* Inability to swallow study medication
* Presence of a medical condition that would make treatment with atomoxetine unsafe (e.g., unstable hypertension or cardiac disease, asthma requiring frequent treatment with albuterol, narrow angle glaucoma, pregnancy, etc.)
* Mental age of less than 18 months
* Previous adequate trial of atomoxetine
* Previous evidence of hypersensitivity or an allergic reaction to atomoxetine
* Clinically significant abnormalities in laboratory measures indicating an undiagnosed medical condition as determined by the study physician in discussion with the participant's primary care physician
* Clinically significant abnormalities on ECG as determined by a pediatric cardiologist
* Pregnant
* Initiation of a new psychosocial intervention within 90 days prior to starting study medication. Participants who have recently had a significant change in their psychosocial interventions will not be eligible until this intervention has been stable for 90 days in order to avoid confounding results of the study. Stable interventions (e.g., speech and occupational therapy) will be allowed to continue during the course of the study. Minor changes in ongoing treatment (e.g., missed therapy sessions due to holiday/vacation planned break in therapy due to school holidays) will not be considered significant.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. McDougle, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Christian Sarkine Autism Treatment Center at Riley Hospital for Children, Indianapolis, Indiana
  - Lurie Center - MassGeneral Hospital, Lexington, Massachusetts

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine (Open Label Trial): Placebo-treated subjects from the randomized trial that don't respond to placebo will be offered an 8-week open-label trial of atomoxetine.
Period: Phase 1-Blinded Randomization (8 weeks)
Arm/Group | Atomoxetine | Placebo | Atomoxetine (Open Label Trial)
Started | 29 | 31 | 0
Completed | 27 | 30 | 0
Not Completed | 2 | 1 | 0
Not completed — no post-baseline ratings | 2 | 1 | 0
Period: Phase 2-Atomoxetine Open Label (8 weeks)
Arm/Group | Atomoxetine | Placebo | Atomoxetine (Open Label Trial)
Started | 0 | 0 | 26
Completed | 0 | 0 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (2.6) | 8.4 (2.1) | 8.8 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 26 | 28 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 22 | 30 | 52
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60
Attending Public School [Count of Participants; unit: Participants] — All children attended school. Children not attending public school attended private, specialized, or home school, or a specialized classroom with type of school unspecified.
  Participants | 24 | 27 | 51
Indiana University School of Medicine Site [Count of Participants; unit: Participants] | 25 | 27 | 52
Tanner Stage 3 or Greater [Count of Participants; unit: Participants] — Tanner stage (1-5) was used to characterize physical development in children, adolescents, and to stratify randomization.The stage was based on external primary and secondary sex characteristics, such as the size of the breasts, genitalia, and development of pubic hair. Tanner stage increases as the child develops. Randomization lists for each of the four strata defined by pubertal status (prepubertal [Tanner Stage I or 2] vs. postpubertal [Tanner Stage 3-5]) and gender (male vs. female) were utilized.
  Participants | 3 | 1 | 4
DSM-IV Diagnosis [Count of Participants; unit: Participants]
  Autistic Disorder | 14 | 9 | 23
  Asperger's Disorder | 5 | 9 | 14
  Pervasive Developmental Disorder (PDD-NOS) | 10 | 13 | 23
Concomitant Medication Use [Count of Participants; unit: Participants] | 22 | 20 | 42
IQ [Mean (Standard Deviation); unit: units on a scale] — IQ was estimated from the Mullen Scale for 1 child assigned to atomoxetine and the Stanford Binet test for all other children. Population: IQ scores were not obtained for 2 children assigned to atomoxetine and 1 child assigned to placebo.
  units on a scale
    number analyzed (Participants) | 27 | 30 | 57
    (all) | 74.7 (18.5) | 84.4 (15.2) | 79.8 (17.4)
Clinical Global Impression-Severity [Count of Participants; unit: Participants]
  Moderate | 16 | 17 | 33
  Marked | 13 | 12 | 25
  Severe | 0 | 2 | 2
Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale Total [Mean (Standard Deviation); unit: units on a scale] — The ADHD Rating Scale (ADHD-RS) is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder with established reliability, validity and sensitivity to change. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). The total score can range from 0 to 54, with a higher score indicating greater severity.
  units on a scale | 37.2 (7.6) | 41.5 (5.8) | 39.4 (7.0)
Aberrant Behavior Checklist, Hyperactivity [Mean (Standard Deviation); unit: units on a scale] | 29.1 (11.8) | 31.7 (10.0) | 30.5 (10.9)
Social Responsiveness Scale [Mean (Standard Deviation); unit: units on a scale] | 84.5 (9.9) | 84.4 (10.3) | 84.5 (10.0)
Vineland Adaptive Behavior Composite Score [Mean (Standard Deviation); unit: units on a scale] — The Vineland Adaptive Behavior Scales, Second Edition is a measure of adaptive behavior in children, adolescents and adults. The composite score has a mean of 100 and a standard deviation of 15 (range = 20 to 160). Higher scores suggest a higher level of adaptive functioning. A rise in standard scores from Baseline to the Final Visit indicates improvement.
  units on a scale | 73.1 (12.5) | 72.5 (8.7) | 72.8 (10.6)
Pediatric Quality of Life Inventory Health Related Functioning [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-100, with higher scores indicating better quality of life.
  units on a scale | 56.3 (18.8) | 60.5 (19.6) | 58.5 (19.2)
Pediatric Quality of Life Inventory Family Functioning [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-100, with higher scores representing better family functioning.
  units on a scale | 52.4 (24.2) | 53.1 (23.4) | 52.7 (23.6)
Pediatric Anxiety Rating Scale, 5-Item Total [Mean (Standard Deviation); unit: units on a scale] — Scaled score ranges form 0-25 with higher scores indicating more severe anxiety symptoms.
  units on a scale | 8.5 (6.5) | 8.9 (6.0) | 8.7 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: ADHD Rating Scale (ADHDRS)-Home Version Total Score (Randomized Phase)
Description: The ADHD Rating Scale (ADHD-RS) is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder with established reliability, validity and sensitivity to change. The ADHD-RS-IV is investigator-administered biweekly during the 8-week double-blind, placebo-controlled phase of the study. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. Results from this rating scale alone should not be used to make a diagnosis. The total score can range form 0 to 54, with a higher score indicating greater severity. Estimates are adjusted for baseline score, study stratum, and site, which were set at their sample means.
Time Frame: 8 weeks
Population: Two participants from the Atomoxetine arm, and one participant from the Placebo arm did not have post-baseline measures.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 27 | 30
units on a scale | 28.7 [24.3 to 33.0] | 34.0 [30.0 to 38.0]

2. Secondary Outcome: ADHD Rating Scale (ADHDRS)-Home Version Inattention and Hyperactivity Scores (Randomized Phase)
Description: The ADHD Rating Scale (ADHD-RS) is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder with established reliability, validity and sensitivity to change. The ADHD-RS-IV is investigator-administered biweekly during the 8-week double-blind, placebo-controlled phase of the study. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. Results from this rating scale alone should not be used to make a diagnosis. The score for each subscale ranges from 0-27 with a higher score indicating greater severity. Estimates are adjusted for baseline score, study stratum, and site, which were set at their sample means.
Time Frame: 8 weeks
Population: Two participants from the Atomoxetine arm, and one participant from the Placebo arm did not have post-baseline measures.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 27 | 30
units on a scale
  Inattention | 14.7 [12.4 to 17.0] | 17.3 [15.2 to 19.4]
  Hyperactivity | 13.7 [11.4 to 16.0] | 16.8 [14.7 to 19.0]

3. Secondary Outcome: Aberrant Behavior Checklist (ABC) (Randomized Phase)
Description: The Aberrant Behavior Checklist (ABC) is a 58-item questionnaire with 5 subscales derived by factor analysis: Irritability, Social Withdrawal, Stereotypy, Hyperactivity, and Inappropriate. It has been extensively used in psychopharmacological studies of autism and assesses many symptoms that are either central to autism (Social Withdrawal, Stereotypy, and Inappropriate Speech) or frequently a target of treatment (Irritability). Each item of the 58-item scale is scored on a 4-point scale (0=never a problem to 3=severe problem). The interpretation of the tool and its sub-scales is that a greater number of items, indicates greater severity. The range of scores per subscale are: Social Withdrawal/Lethargy 0-48; Stereotypy 0-21; Irritability 0-45; Hyperactivity 0-48; Inappropriate Speech 0-12. Parent ratings occur every 2 weeks during the study. Estimates are adjusted for baseline score, study stratum, and site, which were set at their sample means.
Time Frame: 8 weeks
Population: Two participants from the Atomoxetine arm, and one participant from the Placebo arm did not have post-baseline measures.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 27 | 30
units on a scale
  Irritability | 15.6 [12.9 to 18.3] | 13.8 [11.3 to 16.3]
  Lethargy | 7.2 [5.1 to 9.3] | 8.3 [6.3 to 10.2]
  Stereotypy | 4.7 [3.1 to 6.3] | 5.2 [3.7 to 6.6]
  Hyperactivity | 24.2 [20.5 to 27.9] | 28.2 [24.7 to 31.7]
  Inappropriate Speech | 4.4 [3.5 to 5.4] | 5.6 [4.7 to 6.5]

4. Secondary Outcome: Social Responsiveness Scale (SRS) (Randomized Phase)
Description: The Social Responsiveness Scale (SRS) is completed by the parent in order to assess whether additional improvements in social functioning occur with atomoxetine, as observed in our pilot study. This 65-item questionnaire will be completed at baseline and at the end of 8 weeks. The SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each item is summed to create a total score. Total score results as follows: 0-62: within normal limits; 63-79 mild range of impairment; 80-108: moderate range of impairment; 109-149: severe range of impairment. Estimates are adjusted for baseline score, study stratum, and site, which were set at their sample means.
Time Frame: 8 weeks
Population: Four participants from the Atomoxetine arm, and two participants from the Placebo arm did not have post-baseline measures.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale | 83.0 [79.9 to 86.0] | 82.0 [79.2 to 84.8]

5. Secondary Outcome: Vineland Adaptive Behavior Scales (VABS) Composite Score (Randomized Phase)
Description: The Vineland Adaptive Behavior Scales, Second Edition (VABS) is used to assess adaptive functioning in four domains: Communication, Daily Living Skills, Socialization, and Motor Skills. This is a well-standardized open-ended interview used to assess the overall functioning of children and adults. This measure is especially important for subjects with PDDs given that their intellectual level is not always comparable to their adaptive functioning. The Vineland Maladaptive Behavior subscales will be included with these measures as these have been shown to be responsive to drug effects in other clinical trials in this population. The VABS will be done at baseline and at the end of 8 weeks. The composite score represents a standard score (mean = 100 and standard deviation of 15; range = 20-160) on which higher scores indicate a higher level of adaptive functioning. Estimates are adjusted for baseline score, study stratum, and site, which were set at their sample means.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale | 73.4 [70.8 to 76.0] | 74.9 [72.5 to 77.2]

6. Secondary Outcome: Pediatric Quality of Life Inventory (Randomized Phase)
Description: Quality of life is assessed with the Pediatric Quality of Life Inventory (PedsQL 4.0). This instrument is well-validated and widely used for measuring health-related quality of life in children and adolescents. It also appears to be a valid instrument for use with children with psychiatric disorders. The Generic Core scales include 23 items. The health related and family functioning scores range from 0 to 100, with higher scores indicating better quality of life. The Family Impact module will be included to assess any change in family functioning. This will be completed at baseline and at the end of 8 weeks. Estimates are adjusted for baseline score, study stratum, and site, which were set at their sample means.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale
  Health | 64.2 [57.5 to 70.9] | 62.2 [56.0 to 68.4]
  Family | 55.2 [47.3 to 63.0] | 53.0 [45.7 to 60.2]

7. Secondary Outcome: Pediatric Anxiety Rating Scale, 5-Item Total (Randomized Phase)
Description: Since the ABC does not have items which directly assess anxiety, the Pediatric Anxiety Rating Scale (PARS) is administered at week 8 during the study as an exploratory measure. The PARS is a clinician-rated instrument that assesses anxiety symptoms that are commonly associated with social anxiety, separation anxiety, and generalized anxiety disorders. Scaled score ranges form 0-25 with higher scores indicating more severe anxiety symptoms. Estimates are adjusted for baseline score, study stratum, and site, which were set at their sample means.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale | 7.3 [5.6 to 9.1] | 8.5 [6.8 to 10.1]

8. Secondary Outcome: Odds of Clinical Global Impression-Improvement Scale, Very Much or Much Improved (1 or 2) (Randomized Phase)
Description: The Clinical Global Impressions Global Improvement (CGI-I) is designed to take into account all factors to arrive at an assessment of response to treatment. The CGI-I scale ranges from 1 to 7 (1=very much improved; 2= much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse), with lower scores indicating improvement (1=very much improved and 2=much improved). Participants with a CGI-I score of 1 or 2 were classified as improved. Odds of improvement at 8 weeks were estimated using a repeated measures logistic regression model adjusting for baseline severity, study stratum, and site. The CGI-I was administered biweekly during the study. The CGI was focused on the target symptoms of inattention, hyperactivity, and impulsivity.
Time Frame: 8 weeks
Population: Two participants from the Atomoxetine arm, and one participant from the Placebo arm did not have post-baseline measures.
Measure: Number (95% Confidence Interval); unit: odds of improvement
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 27 | 30
odds of improvement | 0.53 [0.22 to 1.26] | 0.11 [0.04 to 0.35]

9. Secondary Outcome: Change in ADHD Rating Scale (ADHDRS)-Home Version Total Score (Open-label Trial)
Description: The ADHD Rating Scale (ADHD-RS) is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder with established reliability, validity and sensitivity to change. The ADHD-RS-IV is investigator-administered biweekly during the 8-week double-blind, placebo-controlled phase of the study. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. Results from this rating scale alone should not be used to make a diagnosis. The total score can range form 0 to 54, with a higher score indicating greater severity. Change will be determined from the start of the open-label trial to 8 weeks post-start.
Time Frame: 8 weeks
Population: Participants randomized to placebo who are not responders at the end of 8 weeks will be treated with atomoxetine for 8 weeks during an open-label trial
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Open-label Trial: Participants randomized to placebo who are not responders at the end of 8 weeks will be treated with atomoxetine for 8 weeks during an open-label trial
Arm/Group | Open-label Trial
Number analyzed (Participants) | 26
units on a scale | -15.4 [-19.9 to -11.0]

10. Secondary Outcome: Change in ADHD Rating Scale (ADHDRS)-Home Version Inattention and Hyperactivity Scores (Open-label Trial)
Description: The ADHD Rating Scale (ADHD-RS) is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder with established reliability, validity and sensitivity to change. The ADHD-RS-IV is investigator-administered biweekly during the 8-week open-label phase of the study. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. Results from this rating scale alone should not be used to make a diagnosis. The score fro each subscale ranges from 0-27, with a higher score indicating greater severity. Change will be determined from the start of the open-label trial to 8 weeks post-start.
Time Frame: 8 weeks
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Trial
Number analyzed (Participants) | 26
units on a scale
  Inattention | -8.1 [-10.4 to -5.7]
  Hyperactivity | -7.3 [-9.7 to -5.0]

11. Secondary Outcome: Change in Aberrant Behavior Checklist (ABC) (Open-label Trial)
Description: The Aberrant Behavior Checklist (ABC) is a 58-item questionnaire with 5 subscales derived by factor analysis: Irritability, Social Withdrawal, Stereotypy, Hyperactivity, and Inappropriate. It has been extensively used in psychopharmacological studies of autism and assesses many symptoms that are either central to autism (Social Withdrawal, Stereotypy, and Inappropriate Speech) or frequently a target of treatment Irritability). Each item of the 58-item scale is scored on a 4-point scale (0=never a problem to 3=severe problem). The interpretation of the tool and its sub-scales is that a greater number of items, indicates greater severity. The range of scores per subscale are: Social Withdrawal/Lethargy 0-48; Stereotypy 0-21; Irritability 0-45; Hyperactivity 0-48; Inappropriate Speech 0-12. Parent ratings occur every 2 weeks during the study. Change will be determined from the start of the open-label trial to 8 weeks post-start.
Time Frame: 8 weeks
Population: Placebo-treated subjects that don't respond to placebo will be offered an 8-week open-label trial of atomoxetine, and the open-label extension will be a continuation phase for those subjects that respond to 8 weeks of atomoxetine during the double-blind phase.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Trial
Number analyzed (Participants) | 26
units on a scale
  Irritability | -4.5 [-7.1 to -1.8]
  Lethargy | -4.0 [-6.1 to -1.9]
  Stereotypy | -2.3 [-3.4 to -1.2]
  Hyperactivity | -11.5 [-15.6 to -7.5]
  Inappropriate Speech | -1.7 [-2.6 to -0.9]

12. Secondary Outcome: Change in Social Responsiveness Scale (SRS) (Open-label Trial)
Description: The Social Responsiveness Scale (SRS) is completed by the parent in order to assess whether additional improvements in social functioning occur with atomoxetine, as observed in our pilot study. This 65-item questionnaire will be completed at baseline and at the end of 8 weeks. The SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each item is summed to create a total score. Total score results as follows: 0-62: within normal limits; 63-79 mild range of impairment; 80-108: moderate range of impairment; 109-149: severe range of impairment. This 65-item questionnaire will be completed at the start of and at the end of 8 weeks of the open-label trial.
Time Frame: 8 weeks
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Trial
Number analyzed (Participants) | 26
units on a scale | -5.8 [-9.5 to -2.1]

13. Secondary Outcome: Change in Vineland Adaptive Behavior Scales (VABS) Composite Score (Open-label Trial)
Description: The Vineland Adaptive Behavior Scales, Second Edition (VABS) is used to assess adaptive functioning in four domains: Communication, Daily Living Skills, Socialization, and Motor Skills. This is a well-standardized open-ended interview used to assess the overall functioning of children and adults. This measure is especially important for subjects with PDDs given that their intellectual level is not always comparable to their adaptive functioning. The Vineland Maladaptive Behavior subscales will be included with these measures as these have been shown to be responsive to drug effects in other clinical trials in this population. The composite score represents a standard score (mean = 100 and standard deviation of 15; range = 20-160) on which higher scores indicate a higher level of adaptive functioning. Change will be determined from the start of the open-label phase to 8 weeks
Time Frame: 8 weeks
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Trial
Number analyzed (Participants) | 26
units on a scale | 5.8 [3.3 to 8.2]

14. Secondary Outcome: Change in Pediatric Quality of Life Inventory (Open-label Trial)
Description: Quality of life is assessed with the Pediatric Quality of Life Inventory (PedsQL 4.0). This instrument is well-validated and widely used for measuring health-related quality of life in children and adolescents. It also appears to be a valid instrument for use with children with psychiatric disorders. The Generic Core scales include 23 items. The health related and family functioning scores range from 0 to 100, with higher scores indicating better quality of life. The Family Impact module will be included to assess any change in family functioning. This will be completed at the start of the open-label trial and at the end of 8 weeks. Change will be determined from the start of the open-label trial to 8 weeks post-start.
Time Frame: 8 weeks
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Trial
Number analyzed (Participants) | 26
units on a scale
  Health | 4.1 [-1.9 to 10.0]
  Family | 13.6 [6.8 to 20.3]

15. Secondary Outcome: Change in Pediatric Anxiety Rating Scale, 5-item Total (Open-label Trial)
Description: Since the ABC does not have items which directly assess anxiety, the Pediatric Anxiety Rating Scale (PARS) is administered at week 8 during the study as an exploratory measure. The PARS is a clinician-rated instrument that assesses anxiety symptoms that are commonly associated with social anxiety, separation anxiety, and generalized anxiety disorders. Scaled score ranges form 0-25 with higher scores indicating more severe anxiety symptoms.Change will be determined from the start of the open-label trial to 8 weeks post-start.
Time Frame: 8 weeks
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Trial
Number analyzed (Participants) | 26
units on a scale | -1.8 [-4.5 to 0.9]

ADVERSE EVENTS:
Groups:
- Atomoxetine (Randomized): Participants will receive flexibly dosed atomoxetine for 8 weeks. Dosage can be increased over the first 4 weeks of study participation and will then be held constant for the remainder of the 8-week trial.
  Atomoxetine: Available tablet strengths of atomoxetine: 5 mg, 10 mg, 25 mg, 40 mg. Week 1 participant takes 0.5 mg/kg/day, Week 2: 0.8 mg/kg/day, Week 3: 1.2 mg/kg/day. Potential exists for dose increase at Week 4 to 1.8 mg/kg/day based on clinical global impression-improvement rating at Week 4.
- Placebo (Randomized): Participants will receive blinded, matched placebo for 8 weeks. Dosage can be increased over the first 4 weeks of study participation and will then be held constant for the remainder of the 8-week trial.
  Placebo: Placebo tablets dosages: 5 mg, 10 mg, 25 mg, 40 mg.
Arm/Group | Atomoxetine (Randomized) | Placebo (Randomized) | Atomoxetine (Open Label Trial)
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31 | 0/26
Other Adverse Events (participants affected / at risk) | 27/29 | 28/31 | 26/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine (Randomized) (N=29) | Placebo (Randomized) (N=31) | Atomoxetine (Open Label Trial) (N=26)
Irritability (Psychiatric disorders) | 10 | 7 | 7
Aggression (Psychiatric disorders) | 5 | 10 | 5
Sedation/drowsiness (General disorders) | 8 | 5 | 8
Headache (Nervous system disorders) | 6 | 6 | 4
Appetite decrease (General disorders) | 9 | 2 | 14
Difficulty falling asleep (Psychiatric disorders) | 6 | 5 | 3
Diarrhea (Gastrointestinal disorders) | 5 | 5 | 4
Self-injurious behavior (Psychiatric disorders) | 6 | 3 | 4
Vomiting (Gastrointestinal disorders) | 5 | 4 | 7
Emotional outburst (Psychiatric disorders) | 5 | 3 | 5
Anxiety (Psychiatric disorders) | 2 | 6 | 1
Increased motor activity (Psychiatric disorders) | 1 | 7 | 2
Change in speech (Psychiatric disorders) | 3 | 4 | 0
Nasal congestion/cold (Infections and infestations) | 4 | 2 | 5
Stomach discomfort (Gastrointestinal disorders) | 4 | 2 | 5
Nightmares or vivid dreams (Psychiatric disorders) | 3 | 3 | 3
Nausea (Gastrointestinal disorders) | 2 | 3 | 4
Fever (General disorders) | 1 | 4 | 1
Social withdrawal (Psychiatric disorders) | 1 | 4 | 2
Restlessness/agitation (Psychiatric disorders) | 4 | 0 | 0
Stereotypy (Psychiatric disorders) | 2 | 2 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Sadness (Psychiatric disorders) | 1 | 3 | 1
Disobedience/defiance (Psychiatric disorders) | 2 | 1 | 1
Flu/upper respiratory (Infections and infestations) | 2 | 1 | 3
Interrupted sleep (Psychiatric disorders) | 2 | 1 | 2
Tiredness/fatigue (General disorders) | 2 | 1 | 1
Disinhibition (Psychiatric disorders) | 1 | 2 | 0
Enuresis (Renal and urinary disorders) | 1 | 2 | 1
Euphoria/giddiness (Psychiatric disorders) | 1 | 2 | 1
Body-focused repetitive behavior (Psychiatric disorders) | 0 | 3 | 0
Not otherwise listed, skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Flushing (Vascular disorders) | 2 | 0 | 0
Appetite increase (General disorders) | 0 | 2 | 0
Accidental injury (General disorders) | 0 | 2 | 0
Eye irritation (Infections and infestations) | 0 | 0 | 2
Sinus condition (Infections and infestations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes